CLINICAL TRIAL: NCT04620096
Title: MENstrual Symptom Tracking to Understand and Assess (Women) Living With Cystic Fibrosis
Acronym: MENSTRUAL
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: University of Illinois at Chicago (Other); University of California, San Diego (Other); Mount Sinai Hospital, New York (Other)
Responsible Party: Principal Investigator, Emily Godfrey, Associate Professor, Department of Family Medicine, University of Washington
Other Study IDs: STUDY00009993; GODFRE20A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2020-10-09; First posted 2020-11-06 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Menstrual Cycle
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystic fibrosis (CF) affects men and women equally, but after the onset of puberty, women with CF have a lower life expectancy than men with CF. Despite these known differences, the link between CF symptom trends and the menstrual cycle remains critically understudied. To address this gap, this study will investigate changes in CF-specific symptoms among women with CF to evaluate whether and how they correlate with their menstrual cycle. Specifically, the investigators hope to examine whether CF-related symptoms change throughout the menstrual cycle, what the impact of those symptoms is on quality of life, and how feasible it is to use a period tracking app to track CF-related symptoms throughout the menstrual cycle. Investigators are asking women ages 18-45 with CF, who have regular menstrual cycles, to participate. Study procedures, including online surveys, period tracking, and interview, will take approximately 3 months.

DETAILED DESCRIPTION:
To better understand the connection between cyclically driven hormone fluctuations and CF-related symptoms, the investigators propose an explanatory, sequential mixed methods study in which 80 menstruating women with CF will be asked to track their daily CF-related symptoms for three consecutive cycles. From this cohort, the investigators will ask up to 30 women with CF to participate in one semi-structured interview to gather information about the impact of cyclical CF symptoms upon women's daily lives and any strategies they use to manage them. This study uses innovative technology to track CF-specific symptoms with a smartphone app. The investigators' hypothesis is that subjective changes in clinical CF symptoms, including pulmonary and sinus (primary outcome), rheumatic, and gastrointestinal (secondary outcomes), will map onto the phases of the menstrual cycle and will be cyclical in nature; women will report alternative ways in which they manage their cyclical CF symptoms; and the period tracker app will be easy for women to use.

ELIGIBILITY:
Inclusion Criteria:

* Females with CF, ages > or = 18 and < 46 years
* Able to read, speak, and understand English
* Have regular menstrual cycles between 21 and 35 days
* If using oral contraceptive pills, patch, or vaginal ring, must have a monthly withdrawal bleed every 21-35 days
* If on a genetic modulator, must be on steady dose for at least 3 months
* Willing to document daily symptoms (or no symptoms) every day for up to four consecutive months
* Has a functioning smartphone app with capability to load a "period tracking" app or, if no smartphone, is willing to complete a paper diary and mail to research team monthly
* Currently resides within the United States

Exclusion Criteria:

* Not regularly menstruating or no regular withdrawal bleed every 21-35 days (with or without hormonal contraception use)
* Planning pregnancy at the start of, or any time during, the 3-month observation period
* Planning to use a hormonal IUD, subdermal contraceptive implant (such as Nexplanon), or injectable contraceptive (such as Depo-Provera) at the start of, or any time during, the 3-month observation period
* Women on the transplant list or what have had a lung transplant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-identify gender as female
Study Population: Regularly menstruating women with Cystic Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Average change of Cystic Fibrosis-related pulmonary symptoms from baseline for each of the four phases of the menstrual cycle (menses, follicular, ovulation, and luteal) | 3 consecutive menstrual cycles (each cycle is 28 days) following enrollment
  Rating of Mild, Moderate, or Severe in the Clue smartphone app
Average change of Cystic Fibrosis-related sinus symptoms from baseline for each of the four phases of the menstrual cycle (menses, follicular, ovulation, and luteal) | 3 consecutive menstrual cycles (each cycle is 28 days) following enrollment
  Rating of Mild, Moderate, or Severe in the Clue smartphone app

SECONDARY OUTCOMES:
Average change of Cystic Fibrosis-related rheumatic symptoms from baseline for each of the four phases of the menstrual cycle (menses, follicular, ovulation, and luteal) | 3 consecutive menstrual cycles (each cycle is 28 days) following enrollment
  Rating of Mild, Moderate, or Severe in the Clue smartphone app
Average change of Cystic Fibrosis-related gastrointestinal symptoms from baseline for each of the four phases of the menstrual cycle (menses, follicular, ovulation, and luteal) | 3 consecutive menstrual cycles (each cycle is 28 days) following enrollment
  Rating of Mild, Moderate, or Severe in the Clue smartphone app

CONTACTS AND LOCATIONS:
Overall Officials: Emily Godfrey, MD, MPH, Principal Investigator — University of Washington; Sandy Sufian, PhD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No